CLINICAL TRIAL: NCT01225601
Title: Epidemiology of Adult Adult Pulmonary Langerhans Cell Histiocytosis - A Multicenter Cohort Study
Brief Title: Prospective Evaluation of Adult Pulmonary Langerhans Cell Histiocytosis
Acronym: LCHA1
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM 04141
Record Dates: First submitted 2010-10-12; First posted 2010-10-21 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2015-03

CONDITIONS: Adult Pulmonary Langerhans Cell Histiocytosis
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Histocytosis: Adult with isolated pulmonary Langerhans cell histiocytosis (pulmonary LCH)
  Interventions: Behavioral: Tabacco discontinuation

INTERVENTIONS:
Behavioral: Tabacco discontinuation — Tabacco discontinuation

SUMMARY:
Study objectives:

* To estimate the incidence of pulmonary deterioration in adult pulmonary Langerhans cell histiocytosis
* To assess the impact of tobacco discontinuation
* Study Design Multicentric prospective cohort study
* Main endpoint: Pulmonary deterioration
* Sample size : 40 patients

DETAILED DESCRIPTION:
Study objectives To estimate the incidence of pulmonary deterioration in adult pulmonary Langerhans cell histiocytosis To assess the impact of tobacco discontinuation Study Design Multicentric prospective cohort study Main endpoint: Pulmonary deterioration Sample size : 40 patients

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary Langerhans cell histiocytosis diagnosed within the past 48 months

Exclusion Criteria:

* Age < 18
* Deep pulmonary dysfunction (CPT< 60%, FEV1< 30%, DLCO< 30%, partial pressure of oxygen in arterial blood (PaO2)< 60mmHg)
* No informed consent or consent withdrawal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Pulmonary Langerhans cell histiocytosis
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2006-05; Primary Completion 2009-05 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Pulmonary deterioration | 2 years
  decrease in Forced expiratory volume in 1 second (FEV1), vital capacity (VC), or Diffusing capacity of the lung for carbon monoxide (DLCO) of at least 15% as compared to baseline values and/or progression of clinical symptoms (general symptoms) and/or occurrence of pneumothorax

SECONDARY OUTCOMES:
Evolution of pulmonary volumes (FEV1) | 6 months
Evolution of pulmonary lesions in High Resolution Computed Tomography (HRCT) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Abdellatif TAZI, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Saint Louis, Paris, Paris, France

REFERENCES:
- [Result] Tazi A, de Margerie C, Naccache JM, Fry S, Dominique S, Jouneau S, Lorillon G, Bugnet E, Chiron R, Wallaert B, Valeyre D, Chevret S. The natural history of adult pulmonary Langerhans cell histiocytosis: a prospective multicentre study. Orphanet J Rare Dis. 2015 Mar 14;10:30. doi: 10.1186/s13023-015-0249-2. PMID 25887097
- [Derived] Tazi A, de Margerie-Mellon C, Vercellino L, Naccache JM, Fry S, Dominique S, Jouneau S, Lorillon G, Bugnet E, Chiron R, Wallaert B, Valeyre D, Chevret S. Extrathoracic investigation in adult patients with isolated pulmonary langerhans cell histiocytosis. Orphanet J Rare Dis. 2016 Feb 2;11:11. doi: 10.1186/s13023-016-0387-1. PMID 26833097